CLINICAL TRIAL: NCT04903353
Title: Pragmatic Trial Comparing Weight Gain in Children With Autism Taking Risperidone Versus Aripiprazole
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Angela Maxwell-Horn, Assistant Professor of Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 210757
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2024-11

CONDITIONS: Weight Gain; Autism Spectrum Disorder; Medication Side Effect
MeSH Terms: conditions — Weight Gain; Autism Spectrum Disorder; Drug-Related Side Effects and Adverse Reactions | interventions — Aripiprazole

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either Risperidone or Aripiprazole after a clinician has chosen to start the patient on an atypical antipsychotic
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment with Risperidone (Active Comparator): Patients prescribed Risperidone
  Interventions: Drug: Comparison of Risperidone and Aripiprazole
- Treatment with Aripiprazole (Active Comparator): Patients prescribed Aripiprazole
  Interventions: Drug: Comparison of Risperidone and Aripiprazole

INTERVENTIONS:
Drug: Comparison of Risperidone and Aripiprazole — Comparing two FDA approved medications for treatment of irritability in autism

SUMMARY:
This study aims to compare two FDA approved medications (aripiprazole and risperidone) for the treatment of behavioral dysregulation in children with autism spectrum disorders. This trial, done in the context of routine clinical care, will seek to evaluate whether aripiprazole or risperidone is associated with more weight gain in children.

DETAILED DESCRIPTION:
Autism is a developmental disability with increasing prevalence in our society. Currently one out of fifty-nine children in the United States has this condition. Many children with autism experience behavioral dysregulation such as irritability and aggression.

Currently, there are two FDA approved atypical antipsychotic medications that treat irritability in children with autism. These are aripiprazole and risperidone. While it is thought that aripiprazole may cause less weight gain than risperidone, clinically this has not been proven.

Understanding the relative risk of ATAP-induced weight gain that results from risperidone versus aripiprazole in a real-world setting could help guide the choice of medical intervention and reduce the cardiometabolic risks, and, most critically, address the limitations of current studies, which have not been able to provide clear clinical insights given the difficulty with having a representative and robust number of patients enrolled.

To be enrolled in this study, participants must be younger than 18 years of age, on the autism spectrum, have behavioral dysregulation, be naive to treatment with atypical antipsychotics and be seen either in the Division of Developmental Medicine or Child and Adolescent Psychiatry at Vanderbilt University Medical Center.

For enrolled patients, the ordering provider will see an order set, randomized to either aripiprazole or risperidone. They will then choose the recommended antipsychotic that the patient has been randomized to, or override the prompt. If the provider overrides the prompt, they will be asked to provide a reason for not choosing the recommended option.

The outcome measure for this study will be weight gain at a 3 month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* age 17 years and younger
* diagnosed with autism
* have behavior problems
* seen in Vanderbilt clinic
* naïve to atypical antipsychotics

Exclusion Criteria:

* 18 years or older
* history of atypical antipsychotic use
* not diagnosed with autism

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 350 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
weight gain | 3 months
  change in weight

CONTACTS AND LOCATIONS:
Overall Officials: Angela Maxwell-Horn, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Division of Developmental Medicine, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No